CLINICAL TRIAL: NCT01609192
Title: Future of Spermatogenesis in Men With Sickle Cell Disease Medically Treated.
Acronym: HYDREP
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: P 081227; AOM 09154 (Other: Assistance Publique)
Record Dates: First submitted 2012-04-25; First posted 2012-05-31 (Estimated); Last update posted 2013-08-07 (Estimated); Status verified 2013-08

CONDITIONS: Drepanocytic Men Treated by Hydroxyurea for the First Time
Keywords: sickle-cell anemia; spermatogenesis; hydroxyurea
MeSH Terms: conditions — Anemia, Sickle Cell | interventions — Hydroxyurea

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- hydroxyurea (Experimental)
  Interventions: Drug: Hydrea® (hydroxyurea )

INTERVENTIONS:
Drug: Hydrea® (hydroxyurea ) — treatment by hydroxyurea (20-30 mg/kg/day) for 6 months

SUMMARY:
The project's background: Sickle cell disease is, at present in France, the most frequent genetic illness. Recent progress in its treatment, in particular the use of hydroxyurea, has considerably modified the prognosis of this disease. Many more patients now reach reproductive age and do consider fathering. Exceptional studies have reported the potential impact of this medical treatment on the sperm parameters and fertility of male patients. In a retrospective analysis, the investigators found that the observed alterations of semen parameters due to sickle cell disease seem to be exacerbated by hydroxyurea treatment.

The study hypothesis: A large prospective study is essential to assess the potential adverse impact of the medical treatment of sickle cell disease on spermatogenesis and consider the advisability of proposing sperm cryopreservation before this treatment is started.

Primary purpose of the protocol: evaluate the impact of a treatment by hydroxyurea (20-30 mg/kg/day), 6 months after its beginning, in 34 men with sickle cell disease (18-60 years old). The main trial criterion will be the average difference of the concentration of spermatozoa s (millions/ml) in the ejaculate, before and after 6 months of medical treatment.

DETAILED DESCRIPTION:
Purpose of the study

Sickle cell disease is, at present in France, the most frequent genetic illness. Recent progress in its treatment, in particular the use of hydroxyurea, has considerably modified the prognosis of this disease. Many more patients now reach reproductive age and do consider fathering. Exceptional studies have reported the potential impact of this medical treatment on the sperm parameters and fertility of male patients. In a retrospective analysis, the investigators found that the observed alterations of semen parameters due to sickle cell disease seem to be exacerbated by hydroxyurea treatment. Moreover, after hydroxyurea cessation, while global results in 30 patients were not statistically different before and after hydroxyurea treatment, in four individuals follow-up sperm parameters did not seem to recover quickly and the total number of spermatozoa per ejaculate fell below the normal range in about half the cases.

Therefore, a large prospective study is essential to assess the potential adverse impact of the medical treatment of sickle cell disease on spermatogenesis and consider the advisability of proposing sperm cryopreservation before this treatment is started.

Main outcomes

Evaluate the impact of a treatment by hydroxyurea (20-30 mg/kg/day), 6 months after its beginning, in 34 men with sickle cell disease (18-60 years old). The primary outcome will be the average difference of the concentration of spermatozoa s (millions/ml) in the ejaculate, before and after 6 months of medical treatment. Six months represent 2 complete cycles of spermatogenesis.

The secondary outcomes will be the other sperm parameters: vitality, mobility, motility, morphology of spermatozoa and the assessment of sperm nuclear DNA fragmentation by TUNEL assay (terminal deoxynucleotidyl transferase dUTP nick end labelling).

This prospective, multicenter, cohort study should allow evaluating the impact of a treatment by hydroxyurea on spermatogenesis in men with sickle cell anemia.

With the hypothesis of a five time reduction in spermatozoa concentration (38 millions ± 43 before treatment), at least 34 analyzable patients are required (aged 18 to 60 years old) who have never received any compound known to be toxic for spermatogenesis.

Protocol

Drepanocytic men who are eligible for a first treatment by hydroxyurea will be sent to the CECOS (center for the study and cryopreservation of oocytes and spermatozoa) at Tenon, Cochin or Jean Verdier hospitals. Their medical history will be recorded and sperm parameters will be analyzed according to WHO criteria. Part of the ejaculate will be fixed and stored (- 20°C) for further DNA fragmentation assay. The rest of the semen could be cryopreserved, according to the patients' will, in case of a potential deleterious effect of the medical treatment on male fertility. Six months after the beginning of the treatment by hydroxyurea, another sperm recovery will be required for the same analysis and the already described parameters will be evaluated and compared to initial results.

Prospects

The study should bring valuable data on the effects of hydroxyurea on human spermatogenesis. If any significant impairment is observed, it would be recommended to perform sperm cryopreservation before the treatment's start.

The study could also help to distinguish between the detrimental effects due to the acute adverse events of sickle cell disease itself and those linked to the administration of hydroxyurea.

ELIGIBILITY:
Inclusion Criteria:

* Men from 18 to 60 years old
* Patients diagnosed with sickle-cell anemia homozygote or S beta thal
* Patients for whom a treatment by hydroxyurea is prescribed for the first time.
* Patients having signed the informed consent
* Patients with social security

Exclusion Criteria:

* Patients already subjected to a treatment potentially sterilizing
* Patients under supervision or guardianship
* Patients that must begin or stop(arrest) a transfusional program between the beginning of the hydroxyurea and the spermogram in 6 months of treatment.
* Rate of ferritin > 2500 µg/l

Ages: 18 Years to 60 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 50 (Actual)
Dates: Start 2010-04; Primary Completion 2013-02 (Actual); Study Completion 2013-02 (Actual)

PRIMARY OUTCOMES:
The primary outcomes will be the average difference of the concentration of spermatozoa in the ejaculate measured before treatment and after 6 months of treatment. | 6 months

SECONDARY OUTCOMES:
the average difference of the sperm DNA fragmentation in the ejaculate measured before treatment and after 6 months of treatment. | 6 months
the average difference of the mobility of spermatozoa in the ejaculate measured before treatment and after 6 months of treatment. | 6 months
the average difference of the vitality of spermatozoa in the ejaculate measured before treatment and after 6 months of treatment. | 6 months
the average difference of the morphology of spermatozoa in the ejaculate measured before treatment and after 6 months of treatment. | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Jacqueline Mandelbaum, Dr, Principal Investigator — Assistance Publique
Locations (1):
- Department of biology of reproduction (TENON Hospital- AP-HP), Paris, France, France